CLINICAL TRIAL: NCT04595981
Title: Chemo-embolization for Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No staff or funding to do the study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jesse G. A. Jones, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006231; UAB (Other: UAB)
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: SCCHN; Squamous Cell Carcinoma
Keywords: Chemo-embolization; Chemoembolization; Squamous Cell Carcinoma of Head and Neck; SCCHN; Platinum-ineligible
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemo-embolization (Experimental): Intra-arterial Cisplatin suspension 150-300 mg is infused into the tumor pedicle(s)
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Subjects will be admitted to the UAB Heart and Vascular Center, pre-medicated with 24 mg Ondansetron IV, 500 mg Prednisolone IV and 1.5 L NaCl with 20 meq KCl IV. The chemo-embolic agent is prepared in the HVC pharmacy by reconstituting 300 mg lyophilized Cisplatin in 60 mL 0.9% NaCl. Subjects are placed under anesthesia in the angiography suite. The access site is prepped and draped in sterile fashion then the femoral artery is catheterized using a 5-French catheter containing a coaxial microcatheter. After superselective visualization of the tumor-feeding vessel, a microcatheter is advanced into the target vessel and infused with 150 mg m2 cisplatin in 45-60 mL NaCl over 30-60 seconds. 10 seconds after the infusion starts, 9 gm sodium thiosulphate is administered IV to neutralize systemic Cisplatin. A post-infusion angiogram is then performed to assess the adequacy of embolization. The catheter is removed and the arteriotomy site closed with a subcutaneous suture.
  Other Names: Platinol

SUMMARY:
The study will evaluate whether adjuvant chemo-embolization increases progression free and/or overall survival relative to standard of care radiation and chemo- and/or immunotherapy in cisplatin-ineligible head and neck cancer patients with an acceptable morbidity rate.

DETAILED DESCRIPTION:
This is a single site, single arm Phase II trial pilot study to explore if chemo-embolization increases progression free and/or overall survival in a subpopulation of cisplatin-ineligible head and neck cancer patients with an acceptable morbidity rate in the U.S. Chemo-embolization will serve as adjuvant therapy performed in addition to standard of care radiation and chemo- and/or immunotherapy. Within UAB, the Investigators plan to recruit 48 patients to implement the intervention, within a two-year period. Progression free survival will be assessed at 3, 6 and 24 months (if available) after intervention, which is determined based upon the results of follow-up Head and Neck imaging (CT or MRI) interpreted by a Radiologist not involved in the study, per standard of care. Overall survival will be reported by the patients' Oncology team on a monthly basis. The trial endpoints will form the basis of how PFS and OS compare to historical outcomes in a similar cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of signed and dated informed consent form
* 2.Stated willingness to comply with all study procedures and availability for the duration of the study
* 3.Male or female, aged 18 or older
* 4.Diagnosed with squamous cell carcinoma of the Head and Neck
* 5.Ability to undergo chemo-embolization
* 6.For females of reproductive potential: Negative pregnancy test at time of chemo-embolization
* 7.Platinum-ineligible as determined by presence of CTS grade I nephropathy, neuropathy or otopathy, and/or ECOG 2+ performance status.
* 8.Plan to undergo standard of care radiation and chemo- and/or immunotherapy.

Exclusion Criteria:

* 1. Medically unfit to undergo chemo-embolization
* 2. Treatment with a competing investigational drug or intervention trial that does not allow adjuvant chemo-embolization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate progression free survival | 6 Months
  Progression free survival is the length of time from the day of the chemo-embolization procedure that a patient lives with the disease but it does not get worse. Cumulative progression-free survival for all patients will be calculated by the Kaplan-Meier method, including the point estimates of progression-free survival and the 95% confidence intervals, evaluated during a six-month period of follow-up.

SECONDARY OUTCOMES:
Evaluate overall survival | 2 Years
  Although the overall survival is related to the primary endpoint (progression free survival), it will be measured independent of the progression free survival. Overall survival is defined for all patients and measured from time of treatment to death or end of a study.
Evaluate oropharyngeal bleeding | 2 years
  Physician visits prompted by new oropharyngeal bleeding that occurs after chemo-embolization will be tabulated. Cumulative bleed-free survival for all patients will be calculated by the Kaplan-Meier method, including the point estimates of bleed-free survival and the 95% confidence intervals, evaluated during a six-month period of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Jones, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No